CLINICAL TRIAL: NCT06006416
Title: Effect of Fenugreek Fibre (Trigonella Foenum-graecum) on the Gut Microbiome in an Adult Population - an Open Label, Self-controlled Trial
Brief Title: Effect of Fenugreek Fibre on Gut Microbiome
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The Sponsor decided not to conduct the study.
Sponsor: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FENGUT
Record Dates: First submitted 2023-08-01; First posted 2023-08-23 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2023-11

CONDITIONS: Gut Microbiome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fenugreek Fibre (Experimental): Fenugreek Fibre - 2 x 10g powder per day with/in food
  Interventions: Drug: Fenugreek Fibre

INTERVENTIONS:
Drug: Fenugreek Fibre — Daily dose of 2 x 10g per day with/in food

SUMMARY:
A open label, self-controlled trial to evaluate the effect of Fenugreek Fibre (Trigonella foenum-graecum) on the gut microbiome in generally healthy adults aged 18-65 years old.

ELIGIBILITY:
Inclusion Criteria:

* Male and females aged 18-65 years old
* Generally healthy
* Able to provide informed consent
* BMI > 25kg/m2
* Agree not to participate in another clinical trial while enrolled in this trial
* Agree not the change their diet or exercise while enrolled in this trial

Exclusion Criteria:

* Unstable(1) or serious illness (e.g. kidney, liver, GIT, heart conditions, diabetes, thyroid gland function, lung conditions, chronic asthma and mood disorders or neurological disorders such as MS)
* Current malignancy (excluding BCC) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years
* Currently taking Coumadin (Warfarin), Heparin, Dalteparin, Enoxaparin or other anticoagulation therapy
* Acute sickness experienced within the past 2 months
* Current use of medications (e.g. antibiotics) or supplements (e.g. pre- and probiotics) that alter the microbiome or gut health. Any use during the trial will result in exclusion from the study.
* Active smokers and/or nicotine or drug abuse
* Chronic alcohol use (>14 alcoholic drinks week)
* Allergic to any of the ingredients in the formula
* Pregnant(2) or lactating woman
* Females of child bearing potential not using a highly effective form of contraception(3,4) (i.e. methods which result in low failure rate, i.e. less than 1% per year, when used consistently and correctly like the oral contraception pill, birth control implant e.g. implanon(3,4))
* People medically prescribed medications that would affect the immune and/or the inflammatory response (e.g. NSAIDs, steroids, antibiotics).
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion
* Participants who have participated in any other related clinical study during the past 1 month
* People with cognitive damage
* People who have or have had treatment for cancer, HIV or chronic use of any dose of steroids (cream, tablet or inhalant) in the past year

Footnotes

1. An unstable illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity. A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments.
2. All female participants of child bearing potential will be required to take a urine pregnancy test prior to entry into the study.
3. Examples of acceptable forms of highly effective contraception include: Established use of oral, injected or implanted hormonal methods of contraception; Placement of an intrauterine device (IUD) or intrauterine system (IUS); Sterilised male partner (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate); True abstinence: When this is in line with your preferred and usual lifestyle
4. Examples of non-acceptable methods of contraception include: Condoms alone or double barrier; Periodic abstinence (e.g. calendar, ovulation, symptothermal, post ovulation); Withdrawal; Spermicide (as it is not approved as a method of contraception in Australia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in metagenomic profile of the gut microbiome | Week 0, week 4 and week 16
  Change in metagenomic profile of the gut microbiome as measured by 16s rRNA gene sequencing

SECONDARY OUTCOMES:
Change in gut function | Week 0, week 4 and week 16
  Change in gut function as measured by faecal short change fatty acids testing via faecal sample
Change in intestinal permeability | Week, 0, week 4, week 8 and week 16
  Change in intestinal permeability as measured by plasma occludin, Muc2 and Endotoxin via blood test
Change in gut inflammation | Week 0, week 4 and week 16
  Change in gut inflammation as measured by faecal calprotectin via faecal sample
Change in inflammation | Week, 0, week 4, week 8 and week 16
  Change in inflammation as measured by inflammatory markers (IFN-g, TNF-a, il-2, MCP-2, IL-1b, TGF-b, CRP) via blood test
Change in GLP-1 | Week, 0, week 4, week 8 and week 16
  Change in GLP-1 as measured by blood test
Change in GST | Week, 0, week 4, week 8 and week 16
  Change in GST as measured by blood test
Change in glutathione | Week, 0, week 4, week 8 and week 16
  Change in glutathione as measured by blood test
Change in FABP | Week, 0, week 4, week 8 and week 16
  Change in FABP as measured by blood test
Change in Homocysteine | Week, 0, week 4, week 8 and week 16
  Change in Homocysteine as measured by blood test
Change in diet | Week 0 and Week 16 (completed for 3 consecutive days)
  Change in diet as measured by 24hr Dietary Recall
Change in quality of life | Week, 0, week 4, week 8 and week 16
  Change in quality of life as measured by the SF-36 questionnaire. Consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Change in stress state | Week, 0, week 4, week 8 and week 16
  Change in stress as measured by the Perceived Stress Scale questionnaire. Consists of 10 items with a score range 0-40. Higher scores indicate higher perceived stress.
Change in sleep quality | Week, 0, week 4, week 8 and week 16
  Change in sleep as measured by the Leeds Sleep Evaluation Questionnaire. Consists of ten questions pertaining to four consecutive aspects of sleep: getting to sleep (GTS), quality of sleep (QOS), awakening from sleep (AFS), and behaviour following wakefulness (BFW). Higher scores indicate better sleep quality.
Change in safety | Week 0, week 4 and week 16
  Change in safety as measured by E/LFT via blood test
Height | Week 0, week 4 and week 16
  Height as measured by stadiometer
Change in weight | Week 0, week 4 and week 16
  Change in weight as measured by digital scale
Change in hip and weight circumference | Week 0, week 4 and week 16
  Change in hip and weight circumference as measured by tape measure
Change in blood pressure | Week 0, week 4 and week 16
  Change in blood pressure as measured by blood pressure monitor

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Rao, PhD, Principal Investigator — RDC Clinical Pty Ltd

IPD SHARING:
Plan to Share IPD: No